CLINICAL TRIAL: NCT07269886
Title: BIOMARKERS FOR DRUG SELECTION IN DEPRESSION: 3BD Test
Brief Title: BIOMARKERS FOR DRUG SELECTION IN DEPRESSION
Acronym: 3BD-Test
Status: Completed | Type: Observational
Sponsor: Neomente SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: Neomente
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- • TAU Group (Treatment as Usual): Patients were followed through standard clinical care.: Patients were evaluated at baseline by the treating physician and subsequently at weeks 8, 12, and 24 by an independent evaluator who was blinded to group allocation.
  The treating physicians of patients in the TAU group received the CDSS information after 12 weeks of follow-up. At that point, they also decided whether or not to consider the CDSS recommendations for pharmacological treatment decisions
- • CDSS Group (Clinical Decision Support Software): The treating physician received CDSS assistance: Psychiatrists received CDSS information and had the option to incorporate it into their treatment decisions starting at T0. Patients were assessed at baseline by the treating psychiatrist and subsequently at weeks 8, 12, and 24 by an independent evaluator who was blinded to group allocation.

SUMMARY:
The study aims to assess whether providing Clinical Decision Support Software (CDSS) information improves the pharmacological response in patients with depression. The CDSS integrates genomic, clinical, and blood biomarker data to assist psychiatrists in selecting the most appropriate treatment for each patient.

A total of 72 patients diagnosed with Major Depressive Disorder were recruited. Participants were male and female adults aged 18 to 65 years, all presenting with moderate to severe symptomatology as assessed by the HAM-D-17 scale.

Enrolled patients were randomized into two groups:

* TAU group (Treatment as Usual) (+): patients received standard clinical care.
* CDSS group: psychiatrists received and could incorporate CDSS-generated information when making treatment decisions.

(+) The TAU group received CDSS information at the 12-week follow-up.

All patients underwent blood collection at baseline (for blood-based and genomic biomarkers) and completed clinical evaluations at baseline, and at 8, 12, and 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Being male or female, aged 18-65.
2. Having a current DSM-5 diagnosis of non-psychotic Major Depressive Disorder confirmed by SCID.
3. Having moderate to severe depressive symptoms as measured by the HAM-D-17.
4. Being indicated for pharmacotherapy for Major Depressive Disorder.
5. Providing written informed consent (signed and dated).

   -

Exclusion Criteria:

1. Having a current or past diagnosis of bipolar disorder or psychotic disorders.
2. Having a moderate to severe substance use disorder within the past six months.
3. Having active suicidal ideation.
4. Having a neurocognitive disorder.
5. Having an unstable or decompensated medical illness likely to confound study outcomes.
6. Being pregnant or lactating.
7. Having known contraindications to the indicated antidepressant classes.
8. Being unable to provide informed consent.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urban depressive outpatients from the City of Buenos Aires were recruited. The population of Buenos Aires is predominantly of Caucasian origin, mainly with ancestry from Italy and Spain.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in depressive symptoms assessed by HAM-D17 | Changes from baseline to week 8
  To evaluate improvement in depressive symptoms after 8 weeks of treatment in the TAU and CDSS groups, assessed by blinded evaluators using the HAM-D17. Change from baseline in HAM-D 17 total score at Week 8 was reported. The HAM-D 17 is a 17-item scale designed to measure the severity of depressive symptoms in participants. Each item reflects a core symptom of major depression. Items are rated on either a 3-point or 5-point scale, with higher scores indicating greater severity. The total score is the sum of all 17 item scores and ranges from 0 to 52, where higher scores indicate greater overall depressive symptom severity. A negative change in score indicates improvement.
  Participant meets response criteria if there is at least a 50% reduction in the HAM-D17 total score from baseline to the last observation carried forward (LOCF) endpoint visit. A participant meets remission criteria if the HAMD-17 total score is less than or equal to 7 at the LOCF endpoint visit.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 items (HAMD-17 | Changes from baseline to week 8 and week 12
  The HAM-D 17 is a 17-item scale. Response is at least a 50% reduction in the 17-item HAM-D17 total score from baseline to the last observation carried forward (LOCF) endpoint visit. Remission is achieved when total score is less than or equal to 7 at the LOCF endpoint visit.
Change in self-administered scale: Patient Health Questionnaire-9 (PHQ-9 | Changes from baseline to week 8 and week 12
  PHQ-9 is a 9 item scale that ranges from 0 to 27 where higher scores indicate higher severity. Response is at least a 50% reduction in the total score from baseline to the LOCF endpoint visit. Remission is achieved when the total score is less than or equal to 4 at the LOCF endpoint visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Neomente, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided